CLINICAL TRIAL: NCT05616221
Title: A Phase 2, Multi-Center, Double-Blind, Randomized, Placebo Controlled Study to Evaluate the Safety, Phage Kinetics, and Efficacy of Inhaled AP-PA02 Multi-Phage Therapeutic in Subjects With Non-Cystic Fibrosis Bronchiectasis and Chronic Pulmonary Pseudomonas Aeruginosa Infection
Brief Title: Study to Evaluate the Safety, Phage Kinetics, and Efficacy of Inhaled AP-PA02 in Subjects With Non-Cystic Fibrosis Bronchiectasis and Chronic Pulmonary Pseudomonas Aeruginosa Infection
Acronym: Tailwind
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP-PA02-201
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Non-cystic Fibrosis Bronchiectasis; Pseudomonas Aeruginosa; Lung Infection
Keywords: Bacteriophage; Phage; NCFB; BE; Pseudomonas; Pseudomonas Aeruginosa
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AP-PA02 (Experimental): Anti-pseudomonal bacteriophage
  Interventions: Biological: AP-PA02
- Placebo (Placebo Comparator): Inactive isotonic solution
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AP-PA02 — Bacteriophage administered via inhalation
  Arms: AP-PA02
Other: Placebo — Inactive Placebo administered via inhalation
  Arms: Placebo

SUMMARY:
A phase 2, multi-center, double-blind, randomized, placebo-controlled study to evaluate the safety, phage kinetics, and efficacy of inhaled AP-PA02 administered in subjects with non-cystic fibrosis bronchiectasis and chronic pulmonary Pseudomonas aeruginosa infection.

DETAILED DESCRIPTION:
This study will be conducted in two cohorts running in parallel: Cohort A will evaluate the safety, tolerability, and efficacy of inhaled AP-PA02 in subjects who have not received an antipseudomonal inhaled antibiotic for a minimum of 3 months prior. Cohort B will evaluate the safety, tolerability, and efficacy of inhaled AP-PA02 in subjects who have received an antipseudomonal inhaled antibiotic for a minimum of 3 months prior. Subjects in both Cohorts A and B will be followed for approximately 4 weeks after last dose of study drug and evaluated for safety, tolerability, and efficacy.

ELIGIBILITY:
Key Inclusion Criteria:

* ≥ 18 years old
* Body mass index (BMI) of ≥ 18 kg/m2
* Evidence of bronchiectasis per CT
* Evidence of chronic pulmonary Pseudomonas aeruginosa infection
* Willing to undergo sputum induction procedures at designated study visits, and willing to provide expectorated sputum samples at all other timepoints (for subjects who are able to expectorate)
* FEV1 ≥ 35% of predicted normal [per Global Lung Function Initiative (GLI) standards] at Screening
* For Cohort A: have not received chronic inhaled antipseudomonal antibiotics regimen for at least 3 months prior to Visit 1
* For Cohort B: have received chronic inhaled antipseudomonal antibiotics regimen for at least 3 months prior to Visit 1

Key Exclusion Criteria:

* Abnormal vital signs at Screening
* History of lung transplantation
* History of cystic fibrosis
* History of α1-antitrypsin deficiency
* History of primary or acquired immunodeficiency syndromes
* History of COPD
* History of pulmonary malignancy or any other malignancy requiring treatment
* History of prolonged QT syndrome
* History of hemoptysis
* Recent significant weight loss
* Recent use of supplemental oxygen during the day while at rest
* Recent use of cigarettes, cigars, or pipes, or used tobacco or other nicotine source by vaping
* Recent changes in either the treatment regimen or initiation of treatment with: oral macrolides, hypertonic saline, mucolytics, bronchodilator medications, or oral corticosteroids
* Currently receiving treatment for active infection at any site
* Female pregnant of breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Velocity Clinical Research, Mobile, Alabama
  - Southern California Institute for Respiratory Diseases Cedars-Sinai West Tower, Los Angeles, California
  - UCONN Health, Farmington, Connecticut
  - Georgetown University Hospital / Pulmonary Critical Care and Sleep Medicine, Washington D.C., District of Columbia
  - Southwest General Healthcare Center, Fort Myers, Florida
  - TecTum Medical Research, Inc., Hollywood, Florida
  - Mayo Clinic/Pulmonary, Critical Care, and Sleep Medicine, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - St. Lukes Hospital, Boise, Idaho
  - The University of Kansas Medical Center / Dept of Medicine, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York Medical College, Hawthorne, New York
  - University of Cincinnati - College of Medicine, Cincinnati, Ohio
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennslyvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - Virginia Commonwealth University (VCU), Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Armata Pharmaceuticals, Inc. — http://armatapharma.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: AP-PA02, 1.5x10^11 PFU/Dose; Cohort A: AP-PA02, 3x10^11 PFU/Dose: Subjects receive AP-PA02
- Cohort A: Placebo: Subjects receive placebo
- Cohort B: AP-PA02, 1.5x10^11 PFU/Dose; Cohort B: AP-PA02, 3x10^11 PFU/Dose: Subjects receive AP-PA02 plus inhaled antibiotic
- Cohort B: Placebo: Subjects receive placebo plus inhaled antibiotic
Period: Overall Study
Arm/Group | Cohort A: AP-PA02, 1.5x10^11 PFU/Dose | Cohort A: AP-PA02, 3x10^11 PFU/Dose | Cohort A: Placebo | Cohort B: AP-PA02, 1.5x10^11 PFU/Dose | Cohort B: AP-PA02, 3x10^11 PFU/Dose | Cohort B: Placebo
Started | 4 | 19 | 12 | 1 | 9 | 3
Completed | 4 | 16 | 12 | 1 | 7 | 3
Not Completed | 0 | 3 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: AP-PA02, 1.5x10^11 PFU/Dose | Cohort A: AP-PA02, 3x10^11 PFU/Dose | Cohort A: Placebo | Cohort B: AP-PA02, 1.5x10^11 PFU/Dose | Cohort B: AP-PA02, 3x10^11 PFU/Dose | Cohort B: Placebo | Total
Number analyzed (Participants) | 4 | 19 | 12 | 1 | 9 | 3 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (7.85) | 60.9 (16.26) | 71.7 (11.02) | 75.0 (0) | 64.1 (16.24) | 53.7 (28.43) | 64.5 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 15 | 8 | 0 | 7 | 3 | 36
  Male | 1 | 4 | 4 | 1 | 2 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 1 | 0 | 3
  White | 3 | 17 | 11 | 0 | 7 | 3 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: P. Aeruginosa Recovery in Sputum Following Multiple Doses of AP-PA02 Administered by Inhalation
Description: Change from baseline in P. Aeruginosa density (colony forming units) as measured in induced sputum samples one week after end of treatment.
Time Frame: Day 17
Population: According to the Statistical Analysis Plan, participants who enrolled before the first DSMB meeting received a lower dose of AP-PA02 (1.5×10¹¹ PFU) and were not included in the primary analysis. In addition, two participants were excluded due to major protocol deviations related to study drug compliance. After applying these prespecified criteria, 41 participants were included in the primary outcome analysis.
Measure: Mean (Standard Deviation); unit: colony forming units log10
Arm/Group | Cohort A: AP-PA02, 1.5x10^11 PFU/Dose | Cohort A: AP-PA02, 3x10^11 PFU/Dose | Cohort A: Placebo | Cohort B: AP-PA02, 1.5x10^11 PFU/Dose | Cohort B: AP-PA02, 3x10^11 PFU/Dose | Cohort B: Placebo
Number analyzed (Participants) | 0 | 18 | 12 | 0 | 8 | 3
colony forming units log10 |  | -0.5 (0.72) | -0.1 (1.11) |  | -0.4 (1.63) | 1.0 (1.13)

2. Post Hoc Outcome: Post Hoc, Pooled Analysis: P. Aeruginosa Recovery in Sputum Following Multiple Doses of AP-PA02 Administered by Inhalation
Description: as for outcome 1
Time Frame: Day 17
Population: Post hoc analysis included all enrolled subjects, regardless of dose level or protocol deviations.
Measure: Mean (Standard Deviation); unit: colony forming units log10
Groups:
- Cohort A + B Pooled AP-PA02: Cohort A + B pooled AP-PA02
- Cohort A + B Pooled Placebo: Cohort A + B pooled placebo
Arm/Group | Cohort A + B Pooled AP-PA02 | Cohort A + B Pooled Placebo
Number analyzed (Participants) | 33 | 15
colony forming units log10 | -0.6 (0.93) | 0.1 (1.17)

ADVERSE EVENTS:
Time Frame: 38 Days
Arm/Group | Cohort A: AP-PA02, 1.5x10^11 PFU/Dose | Cohort A: AP-PA02, 3x10^11 PFU/Dose | Cohort A: Placebo | Cohort B: AP-PA02, 1.5x10^11 PFU/Dose | Cohort B: AP-PA02, 3x10^11 PFU/Dose | Cohort B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/19 | 0/12 | 0/1 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/19 | 0/12 | 0/1 | 3/9 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 15/19 | 5/12 | 0/1 | 7/9 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: AP-PA02, 1.5x10^11 PFU/Dose (N=4) | Cohort A: AP-PA02, 3x10^11 PFU/Dose (N=19) | Cohort A: Placebo (N=12) | Cohort B: AP-PA02, 1.5x10^11 PFU/Dose (N=1) | Cohort B: AP-PA02, 3x10^11 PFU/Dose (N=9) | Cohort B: Placebo (N=3)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: AP-PA02, 1.5x10^11 PFU/Dose (N=4) | Cohort A: AP-PA02, 3x10^11 PFU/Dose (N=19) | Cohort A: Placebo (N=12) | Cohort B: AP-PA02, 1.5x10^11 PFU/Dose (N=1) | Cohort B: AP-PA02, 3x10^11 PFU/Dose (N=9) | Cohort B: Placebo (N=3)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum purulent (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulation time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT05616221/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT05616221/SAP_001.pdf